CLINICAL TRIAL: NCT04408820
Title: Specified Drug Use-Results Survey of EVRENZO® Tablets: Non-interventional, Prospective Drug Use-results Survey in the Realworld Use of EVRENZO® Tablets (Roxadustat) in Patients With Renal Anemia
Brief Title: Post-marketing Surveillance of EVRENZO® Tablets (Roxadustat) in Patients With Renal Anemia
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 1517-MA-3318
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Renal Anemia
Keywords: ASP1517; Evrenzo; Roxadustat
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Roxadustat: Participants will receive oral dose of roxadustat.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Oral
  Other Names: ASP1517; Evrenzo

SUMMARY:
The purpose of this study is to assess the safety and efficacy, including the incidence of thromboembolism, in renal anemia patients treated with roxadustat (EVRENZO® Tablets) in actual clinical settings.

DETAILED DESCRIPTION:
This is a post-marketing long-term specified drug use-result survey study required for products in Japan. In the survey, patient registration and data collection will be conducted using post-marketing survey data collection system, PostMaNet via the Internet.

Patients who are eligible for the survey will be registered within 14 days after the start of treatment with roxadustat (including the start day of treatment). For all registered patients (including discontinuations/dropouts), the investigator will enter the necessary information in the case report form (CRF) and send it immediately after the end of the specified observation period for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Renal anemia patients who are naïve to roxadustat.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Renal anemia patients on dialysis and non-dialysis who are naïve to roxadustat
Sampling Method: Non-Probability Sample
Enrollment: 2104 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Adverse Drug Reactions (ADR) | Up to Week 104
  An AE is defined as any unwanted medical occurrence after drug administration and which does not necessarily have a causal relationship with the treatment.
  ADR is AEs whose relationship to the study drugs could not be ruled out is considered adverse drug reaction. AEs that fall under either "Probable" or "Possible" or "Unassessable" should be defined as "AEs whose relationship to the study drugs could not be ruled out.
Proportion of participants with serious ADR | Up to Week 104
  ADR is considered "serious" if, in the view of the investigator, the event: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires hospitalization or prolongation to hospitalization, or other medically important event.
Proportion of participants with thromboembolism | Up to Week 104
  Number of participants with thromboembolism compared to number of participants evaluated.
Proportion of participants with hypertension | Up to Week 104
  Number of participants with hypertension compared to number of participants evaluated.
Proportion of participants with hepatic function disorder | Up to Week 104
  Number of participants with hepatic function disorder compared to number of participants evaluated.
Proportion of participants with malignant tumors | Up to Week 104
  Number of participants with malignant tumors compared to number of participants evaluated.
Proportion of participants with retinal hemorrhage | Up to Week 104
  Number of participants with retinal hemorrhage compared to number of participants evaluated.
Proportion of Participants With Seizures | Up to week 104
  Number of participants with seizures will be reported.
Proportion of Participants With Serious Infection | Up to week 104
  Number of participants with serious infection will be reported.
Proportion of Participants With Central Hypothyroidsm | Up to Week 104
  Number of participants with central hypothyroidsm compared to number of participants evaluated.
Proportion of participants with myopathy events | Up to Week 104
  Number of participants with myopathy events related to the concomitant use of hydroxymethylglutaryl-CoA (HMG-CoA) reductase inhibitors compared to number of participants evaluated.
Proportion of Participants With Renal Function Disorder | Up to week 104
  Number of participants with renal function disorder reported as adverse drug reaction in participants with autosomal dominant polycystic kidney disease (ADPKD) will be reported.
Proportion of participants with ADR within 4 weeks after switching to roxadustat | Up to Week 4
  Number of participants with ADR within 4 weeks after switching from erythropoiesis stimulating agent (ESA) to roxadustat compared to number of participants evaluated.
Proportion of participants with ADR with high doses of roxadustat | Up to Week 104
  Number of participants with ADR with high doses of roxadustat compared to number of participants evaluated.
Change from baseline in Hemoglobin (Hb) levels | Up to Week 104
  Hb will be recorded from blood samples collected.
Mean value of Hb levels over time | Up to Week 104
  Hb will be measured throughout the period.
Achievement rate for target Hb level | Up to Week 104
  Percent of participants who achieved target Hb level (10.0 to 12.0 g/dL).
Mean Hb levels at 4 weeks after switching to roxadustat | At Week 4
  Hb levels at 4 weeks after switching from ESA to roxadustat.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Inc., Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00023, Aichi
  - Site JP00005, Akita
  - Site JP00002, Aomori
  - Site JP00012, Chiba
  - Site JP00038, Ehime
  - Site JP00018, Fukui
  - Site JP00040, Fukuoka
  - Site JP00007, Fukushima
  - Site JP00021, Gifu
  - Site JP00010, Gunma
  - Site JP00034, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00028, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00017, Ishikawa
  - Site JP00037, Kagawa
  - Site JP00046, Kagoshima
  - Site JP00014, Kanagawa
  - Site JP00039, Kochi
  - Site JP00043, Kumamoto
  - Site JP00026, Kyoto
  - Site JP00024, Mie
  - Site JP00004, Miyagi
  - Site JP00045, Miyazaki
  - Site JP00020, Nagano
  - Site JP00042, Nagasaki
  - Site JP00029, Nara
  - Site JP00015, Niigata
  - Site JP00003, Numakunai
  - Site JP00033, Okayama
  - Site JP00047, Okinawa
  - Site JP00027, Osaka
  - Site JP00044, Ōita
  - Site JP00041, Saga
  - Site JP00011, Saitama
  - Site JP00025, Shiga
  - Site JP00032, Shimane
  - Site JP00022, Shizuoka
  - Site JP00009, Tochigi
  - Site JP00036, Tokushima
  - Site JP00013, Tokyo
  - Site JP00031, Tottori
  - Site JP00016, Toyama
  - Site JP00030, Wakayama
  - Site JP00006, Yamagata
  - Site JP00035, Yamaguchi
  - Site JP00019, Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tsuruya K, Sugamori H, Tanaka Y, Wakasugi N, Ito Y. Real-world safety and effectiveness of roxadustat in patients with anemia of chronic kidney disease: interim results from a post-marketing surveillance study in Japan. Expert Opin Pharmacother. 2025 Mar;26(4):503-517. doi: 10.1080/14656566.2025.2462181. Epub 2025 Feb 7. PMID 39899733